CLINICAL TRIAL: NCT06912061
Title: A Needle Technique for Achilles Tendon Lengthening in Pediatric Patients: A Prospective Study on Efficacy, Safety, and Feasibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 703025
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Equinus Contracture
Keywords: Idiopathic toe walking (ITW); Tendon Achilles Lengthening (TAL); needle technique
MeSH Terms: conditions — Equinus Deformity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tendon Achilles Lengthening using needle technique (Active Comparator): The arm in question involves the administration of a specific intervention via a precise needle technique, as outlined in the study protocol. The needle technique employed ensures optimal delivery of the intervention, ensuring safety and efficacy for the patient population under investigation. Further details regarding the needle technique are described in the full protocol.
  Interventions: Procedure: Needle tendon lengthening technique

INTERVENTIONS:
Procedure: Needle tendon lengthening technique — Percutaneous Achilles tendon lengthening with the needle technique is performed by applying a series of microtenotomies to the tendon using needle pricks while the tendon is stretched. A withdrawal needle with a diameter of 1.1-1.2 mm is used. The needle pricks gradually weaken the tendon and stretch it to the desired length without opening the skin or tendon sheath. As a rule, it is desirable to achieve approximately 10-15 degrees of dorsiflexion before concluding the lengthening.
  Local infiltration anesthesia is applied, followed by a simple bandage. The surgical procedure typically takes 3-4 minutes. Finally, a boot cast in soft plaster with the foot and ankle in neutral position is applied, and it can be fully weight-bearing immediately.
  The cast is removed at the clinic after 4 weeks. After cast removal, the child/adolescent should be allowed gentle activity - not sports - for another 4 weeks, thereafter unrestricted activity.
  Physical therapy may be utilized as needed, locally.

SUMMARY:
For years, we have used a minimally invasive and biological variant of Achilles tendon lengthening using a needle inserted into the Achilles tendon so that it is weakened and can be gradually stretched to the desired length. So far, no negative effects, complications or tendon problems have been observed. A prospective study of a cohort of children and adolescents is planned where there is an indication for Achilles lengthening, such as spastic or non-spastic contracture and toe walking that results in an unwanted shortening of the Achilles tendon that makes walking difficult. We plan to include up to 50 children and adolescents over a two-year period and follow them closely for the first year after surgery. Pediatric physiotherapists will perform all clinical examinations to limit observer bias, and a radiologist will examine the tendon tissue with ultrasound before and one year after surgery to check anatomical conditions. The study will examine safety, effectiveness and feasibility of using the method, and anatomy, patient satisfaction and quality of life.

DETAILED DESCRIPTION:
cases of restriction. Traditionally, Achilles tendon lengthening has been performed through open surgery using Z lengthening or sliding techniques, or percutaneously with 2-3 partial cuts using a scalpel. However, these methods may lead to scarring and other complications that some find troublesome.

A novel technique for Achilles tendon lengthening involves the needle technique, which applies a series of percutaneous microtenotomies to the tendon using needle pricks. These microtenotomies gradually weaken and stretch the tendon to the desired length without necessitating the opening of the skin or tendon sheath, thus avoiding scar formation. This modified technique may offer potential advantages over traditional methods, yet there is limited research in this area. It is also unknown how the Achilles tendon reorganizes anatomically following needle lengthening. The technique is similar to that used in the percutaneous release of Dupuytren's contracture, and several reports have emerged on the use of this method for Achilles tenotomy in the treatment of clubfoot. Ultrasound-guided needle techniques for gastrocnemius recession have also been reported. We have utilized this technique in approximately 200 patients over the past few years with positive experiences, both in terms of surgical technique and clinical outcomes. Patients predominantly report positive experiences with significant benefits from the lengthening.

The purpose of this study is to evaluate the needle technique as a surgical method for Achilles tendon lengthening in children and adolescents. The study will assess the efficacy, feasibility, and safety of the percutaneous needle technique for Achilles tendon lengthening in pediatric patients. The study aims to contribute to the knowledge of a new and likely more benign surgical method for treating equinus foot deformities in children and to evaluate whether the needle technique can be a safe, effective, and feasible alternative to existing treatments.

Objective:

To compare the efficacy and safety of two surgical techniques (needle technique vs. standard Z-plasty) for Achilles tendon lengthening in pediatric patients aged ≥ 5 to ≤ 16 years.

Study Design:

A prospective observation of a cohort of young patients undergoing Achilles tendon lengthening using the needle technique over a two-year period.

Sample Size:

Up to 50 patients will be recruited, or as many as consent to participate during the two-year study period. No significant differences regarding the effect of the procedure are expected. Since the occurrence of complications following this type of surgery is very rare, the sample size is determined at discretion. A sample size based on statistical calculations to ensure the study's ability to detect meaningful differences in the study group compared to historical findings would necessitate an impractically large group of patients.

Methods

Procedure:

Percutaneous Achilles tendon lengthening with the needle technique is performed by applying a series of microtenotomies to the tendon using needle pricks while the tendon is stretched. A withdrawal needle with a diameter of 1.1-1.2 mm is used. The needle pricks gradually weaken the tendon and stretch it to the desired length without opening the skin or tendon sheath. As a rule, it is desirable to achieve approximately 10-15 degrees of dorsiflexion before concluding the lengthening.

Local infiltration anesthesia is applied, followed by a simple bandage. The surgical procedure typically takes 3-4 minutes. Finally, a boot cast in soft plaster with the foot and ankle in neutral position is applied, and it can be fully weight-bearing immediately.

The cast is removed at the clinic after 4 weeks. After cast removal, the child/adolescent should be allowed gentle activity - not sports - for another 4 weeks, thereafter unrestricted activity.

Physical therapy may be utilized as needed, locally. Radiology Routine conventional radiographs of the feet/ankles are not taken. Ultrasound examination is conducted just before and one year after the procedure.

Ultrasound Method: Use of a high-frequency linear transducer for accurate assessment of the Achilles tendon.

Clinical Examination The tests and measurements are standardized and conducted by two experienced testers (pediatric physiotherapists) using a goniometer. The patients are lying on a bench during the examination. In cases of doubt or uncertain measurements, the examinations are repeated as many times as necessary and the average is used. Strength testing is performed before and one year after the operation with a handheld dynamometer.

An orienting neurological examination, i.e., assessment of spasticity (MAS), reflex Preliminary Neurological Examination, i.e., assessment of spasticity (MAS), reflexes, clonus, is performed prior to the surgery to uncover any underlying neurological condition.

Quality of Life A validated translated version of the generic PedsQL scale will be used to assess the patients' HRQoL, based on age (18-20). Self-reports will be used for patients aged 5-7, 8-12, and 13-18 years. Parent-proxy reports will be used for the ages of 5-7, 8-12, and 13-18. Parents will complete the parent-proxy report independently from the patient and in separate rooms. PedsQL score reports will be completed during preoperative and 1-year follow-up assessments.

Data Collection:

Data will be collected before the procedure, and at 4 weeks, 6 months, and one year after the procedure at specified follow-up intervals. Standardized forms for data collection will be used to ensure uniformity in data collection.

Statistical Analysis:

Paired t-tests will be used for comparison of continuous and normally distributed data. Fisher's exact test will be used for comparison of dichotomous parameters. SPSS 28 will be used for data analysis, and a p-value <0.05 will be considered statistically significant.

Project Organization and Data Storage:

The study is conducted by the project group at the Department of Orthopedics, Drammen Hospital. The project group holds the data necessary for the study and owns the data. Nettskjema is used for data collection, and the data are stored on Medinsight on a secure research server. During the study, indirectly identifiable information is stored on the research server in the Research Portal for HSØ, where all project participants have access. The code list is stored separately from these and locked in a secure, locked cabinet (safe).

Ethics and Consent:

The study will be conducted in accordance with the Helsinki Declaration and local ethical guidelines. Applications will be made to the Regional Committees for Medical and Health Research Ethics (REK) and the Data Protection Officer (PVO) in VV. Informed consent for participation, data use, and publication permission will be obtained from parents/guardians (all participants are under 16 years), and information letters will be prepared and distributed to the children according to age (5-12, 12-16).

See attached consent form.

Study Registration:

The study will be registered in a recognized clinical study registry to ensure transparency.

Patient recruitment is planned to start in the fall of 2024. A 2-year inclusion period is estimated, meaning inclusion is expected to be completed by the fall of 2026. If necessary, an extension of the study period will be requested from REK and PVO. Data collection at follow-up, etc., is estimated to be completed by the fall of 2027.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5-16 years
* Consent from parents/guardians
* Indication for Achilles tendon lengthening (toe walking, spasticity), both unilateral and bilateral:
* Equinus foot with dorsiflexion ≤ 0 degrees with the knee extended and the heel in neutral position.
* Symptomatic equinus foot, meaning a foot position causing pain, discomfort, increased fatigue, etc.

Exclusion Criteria:

* Unwillingness to participate, lack of consent
* Previous surgical Achilles tendon lengthening, e.g., for clubfoot
* Received BoNT-a injection in the triceps surae within the last 6 months
* Contracture in the ankle joint, i.e., equinus position not due to a tight Achilles tendon
* Positive Silfverskiöld test and dorsiflexion > 5 degrees with the knee extended (indicating the need for gastrocnemius recession)
* Concurrent other surgery/other procedures on the same lower extremity, including BoNT-a injection

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Passive ankle dorsiflexion (PDF) | Baseline, as measured preoperatively, then after 4 weeks, 6 months, and one year after the surgery.
  Passive ankle dorsiflexion (PDF) (degrees) lying down with an extended knee using a goniometer. The examination is performed by experienced physiotherapists that are not involved in the project.

SECONDARY OUTCOMES:
Passive ankle dorsiflexion (PDF) | Baseline, as measured preoperatively, then after 4 weeks, 6 months, and one year after surgery.
  Passive ankle dorsiflexion (PDF) (degrees) with a bent knee using a goniometer. The examination is performed by experienced physiotherapists that are not involved in the project.
Active ankle dorsiflexion (ADF) | Baseline, as measured preoperatively, then after 4 weeks, 6 months, and one year after the surgery.
  Active ankle dorsiflexion (ADF) (degrees) with a bent knee (goniometer). The examination is performed by experienced physiotherapists that are not involved in the project.
Plantar flexion strength | Baseline, as measured preoperatively, then after 6 months, and one year after the surgery.
  Plantar flexion strength (Kg) as measured clinically and with a handheld dynamometer, performed by experienced physiotherapists that are not involved in the science project.
Complications and adverse events | At follow-up check-ups after 4 weeks, 6 months, and one year after the surgery.
  All complications and adverse events, such as re-ruptures, wound infections, bleeding, and necrosis within the first postoperative year are noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Drammen Sykehus, Vestre Viken HF, Drammen, Norway

IPD SHARING:
Plan to Share IPD: No
Sharing data is prohibited by the Ethics Committee, both the Regional Committee (REK) and the local Patient Protection Committee (PVO)